CLINICAL TRIAL: NCT01418339
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Flexible-Dose Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Brief Title: Efficacy & Safety Study of Once-weekly Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-10-272; 2011-000467-27 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-17 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Tourette's Disorder
Keywords: Tourette's Disorder; Tic disorders
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aripiprazole (Experimental): Aripiprazole was administered orally once a week (QW) for 8 weeks in a double-blind manner. Participants randomized to aripiprazole received aripiprazole tablets at a starting dose of 52.5 milligrams (mg) QW on Day 0. At Week 1, according to the investigator's discretion based on efficacy and tolerability, the dose of aripiprazole could remain at 52.5 mg QW or could be increased to 77.5 mg QW. The dose could be increased to 110 mg QW as early as Week 2. For the remainder of the study (up to Week 8), the dose was to be adjusted up and down among these three dose levels, as determined by the investigator.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Participants randomized to placebo received aripiprazole-matching placebo, tablet, orally, QW for 8 weeks in a double-blind manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole tablet administered orally once a week.
  Other Names: ABILIFY
  Arms: Aripiprazole
Drug: Placebo — Aripiprazole-matching placebo tablet administered orally once a week.
  Arms: Placebo

SUMMARY:
The goal of the current study is to determine efficacy and safety of once-weekly aripiprazole in reducing Total Tic Severity (TTS) score in children and adolescents with Tourette's Disorder.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 17 year old with diagnostic and statistical manual of mental disorders, fourth edition -text revision (DSM-IV-TR) diagnostic criteria for Tourette's disorder (TD), confirmed by the kiddie schedule for affective disorders and schizophrenia - present and lifetime version (K-SADS-PL), including the Diagnostic Supplement 5
* Has a total tic score (TTS) ≥20 on the yale global tic severity scale (YGTSS) at Screening and Baseline
* Presenting tic symptoms cause impairment in the participant's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships
* Females of childbearing potential must have a negative pregnancy test, must be practicing acceptable double-barrier methods of contraception, and must not be pregnant or lactating.
* Written informed consent form (ICF) obtained from a legally acceptable representative & informed assent at Screening as applicable by study center's Institutional review board/independent ethics committee (IRB/IEC)
* The participant, designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator.

Exclusion Criteria:

* Clinical presentation and/or history, consistent with another neurologic condition that may have accompanying abnormal movements.
* History of schizophrenia, bipolar disorder, or other psychotic disorder.
* Participant receiving psychostimulants for treatment of attention-deficit disorder/Attention-deficit hyperactivity disorder (ADD/ADHD) and who have developed and/or had exacerbations of tic disorder after initiation of stimulant treatment.
* Currently meets DSM-IV-TR criteria for a primary mood disorder.
* Severe obsessive-compulsive disorder (OCD), per children's yale-brown obsessive compulsive scale (CY-BOCS) score >16.
* Taken aripiprazole within 30 days of the Screening visit.
* Received any investigational agent in a clinical trial within 30 days prior to Screening or who were randomized into a clinical trial with Once-weekly aripiprazole at any time.
* History of neuroleptic malignant syndrome.
* Sexually active participants not using 2 approved methods of contraception; breastfeeding or pregnant.
* Risk of committing suicide
* Bodyweight lower than 16 kg
* Taken neuroleptic or antiparkinson drugs <14 days prior to randomization.
* Requiring cognitive-behavioral therapy (CBT) for TD during study.
* Participant meets DSM-IV-TR criteria for any significant psychoactive substance use disorder within the past 3 months.
* Positive drug screen
* Participant requires medications not allowed per protocol
* Use of CYP2D6 and CYP3A4 inhibitors or CYP3A4 inducers within 14 days prior to dosing and for duration of study.
* Inability to swallow tablets or tolerate oral medication
* Abnormal laboratory test results, vital signs and Electrocardiogram (ECG) results

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2011-07-27 (Actual); Primary Completion 2013-11-06 (Actual); Study Completion 2013-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (35):
- United States (19):
  - Little Rock, Arkansas
  - Sacramento, California
  - Santa Ana, California
  - Wildomar, California
  - Hialeah, Florida
  - Orange City, Florida
  - St. Petersburg, Florida
  - Overland Park, Kansas
  - New Orleans, Louisiana
  - Bloomfield Hills, Michigan
  - Staten Island, New York
  - Avon Lake, Ohio
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Bothell, Washington
- Canada (3):
  - Kelowna, British Columbia
  - Toronto, Ontario
  - Whitby, Ontario
- Hungary (2):
  - Budapest
  - Szeged
- Mexico (3):
  - León, Guanajuato
  - Monterrey, Nuevo León
  - Durango
- South Korea (4):
  - Gyeonggi-do
  - Gyeongsang
  - Incheon
  - Seoul
- Taiwan (4):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/.
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 152 participants were screened and 135 were randomized to the treatment. The randomized participants were recruited from 45 study sites in the following 6 countries: United States (US), Hungary, Canada, Taiwan, South Korea, and Mexico. Out of 135, 124 participants were included in the modified intention-to-treat (mITT) population.
Pre-assignment Details: The study consisted of a Pretreatment and Treatment Phase. The Pretreatment Phase consisted of a Screening Period, Washout Period (when applicable), and Baseline visit. This was followed by an 8-week Treatment Phase. There was also a Follow-up Period (30 days) for participants who did not roll over into the open-label study 31-10-274 (NCT01416441).
Groups:
- Placebo: Participants randomized to placebo received aripiprazole-matching placebo tablet, orally, QW for 8 weeks in a double-blind manner.
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 90 | 45
Completed | 78 | 35
Not Completed | 12 | 10
Not completed — Adverse Event | 5 | 2
Not completed — Subject Withdrew Consent | 1 | 2
Not completed — Lack of Efficacy as Determined by the Investigator | 6 | 6

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) included all participants randomly assigned to the double-blind treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 90 | 45 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.9 (2.8) | 11.7 (2.6) | 11.9 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 73 | 31 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 13 | 33
  Not Hispanic or Latino | 67 | 31 | 98
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 28 | 12 | 40
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 1 | 4
  White | 53 | 31 | 84
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Yale Global Tic Severity Scale (YGTSS) -Total Tic Score (TTS) [Mean (Standard Deviation); unit: score on a scale] — The YGTSS is a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The total tic score (TTS) ranged from 0 (none) to 50 (severe) with higher score represent more severe symptoms.
  score on a scale | 30.5 (6.6) | 29.3 (7.0) | 30.1 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Yale Global Tic Severity Scale (YGTSS) - Total Tic Score (TTS)
Description: The YGTSS is a semi-structured clinical interview designed to measure the tic severity. This scale consisted of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings were made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics, each including number, frequency, intensity, complexity, and interference. The YGTSS TTS was the summation of the severity scores of motor and vocal tics. The TTS ranged from 0 (none) to 50 (severe) with a higher score represent more severe symptoms (greater reduction from baseline for greater improvement). Mixed Effect Repeated Measure Model (MMRM) analysis was performed.
Time Frame: Baseline to Week 8
Population: Modified Intention-to-Treat (mITT) included all participants randomly assigned to the double-blind treatment, excluding participants from the two sites that were terminated. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 71 | 34
score on a scale | -12.34 (0.88) | -7.72 (1.23)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; The statistical comparison was performed using MMRM model at a significance level of 0.05 (2-sided); Test type: Superiority; p = 0.0028, MMRM — P-value was derived from a repeated measures linear model with treatment, week, and treatment by week interaction as fixed categorical effects, the baseline value as a fixed covariate, and week as the time variable for repeated measures; Treatment Difference = -4.63, 95% CI 2-sided [-7.62 to -1.63]

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions Scale for Tourette's Syndrome (CGI-TS) Score
Description: The severity of illness and efficacy of study medication for each participant were rated using the CGI-TS scale. The study physician rated the participants total improvement whether or not it is due to study treatment. All responses were compared to the participants condition at Baseline (Day 0). Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients), with lower score indicating better improvement. A negative change from Baseline indicates improvement. MMRM analysis was performed.
Time Frame: Baseline to Week 8
Population: mITT included all participants randomly assigned to the double-blind treatment, excluding participants from the two sites that were terminated. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 70 | 33
score on a scale | 2.29 (0.12) | 2.81 (0.17)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; The statistical comparison was performed using MMRM model at a significance level of 0.05 (2-sided); Test type: Superiority; p = 0.0124, MMRM — [p-value comment as in outcome 1, analysis 1]; Treatment Difference = -0.52, 95% CI 2-sided [-0.93 to -0.12]

3. Secondary Outcome: Change From Baseline in Gilles de la Tourette Syndrome - Quality of Life Scale (GTS-QOL) Total Score
Description: The GTS-QOL is a disease-specific patient-reported scale for the measurement of health-related quality of life in participants with Tourette's Disorder, taking into account the complexity of the clinical picture of the disease. The questionnaire consists of a 27-item Tourette's Disorder-specific scale with 4 subscales (psychological, physical, obsessional, and cognitive). The GTS-QOL total score ranged from 0 (extremely dissatisfied with life) and 100 (extremely satisfied with life). A positive change from Baseline indicates improvement. MMRM analysis was performed.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 71 | 34
score on a scale | 10.04 (1.83) | 12.04 (2.60)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; The statistical comparison was performed using MMRM model at a significance level of 0.05 (2-sided); Test type: Superiority; p = 0.5317, MMRM — [p-value comment as in outcome 1, analysis 1]; Treatment Difference = -2.00, 95% CI 2-sided [-8.31 to 4.32]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose (Up to approximately 12 weeks)
Description: Safety Sample included all participants in the ITT Sample who received at least 1 dose of study drug.
Arm/Group | Aripiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/90 | 0/45
Other Adverse Events (participants affected / at risk) | 38/90 | 8/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=90) | Placebo (N=45)
Hyperthermia (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Dystonia (Nervous system disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=90) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 12 | 4
Vomiting (Gastrointestinal disorders) | 9 | 1
Fatigue (General disorders) | 8 | 0
Increased Appetite (Metabolism and nutrition disorders) | 6 | 1
Headache (Nervous system disorders) | 12 | 2
Somnolence (Nervous system disorders) | 15 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.